CLINICAL TRIAL: NCT02186899
Title: Comparison of Femoral - Sciatic - Obturator Nerve Block vs General Anesthesia in Combination With Continuous or Bolus Femoral Nerve Block for Arthroscopic ACL Repair Regarding the Time of Patient Mobilasation
Brief Title: Peripheral Nerve Block (Femoral - Sciatic - Obturator) Versus General Anesthesia for Arthroscopic ACL Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Marina Simaioforidou, Anesthesiologist, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FSOvsGA
Record Dates: First submitted 2014-04-27; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Arthroscopic ACL Rerpair; Surgery; Anesthesia Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- General Anesthesia Femoral continuous (Active Comparator): General anesthesia plus continuous femoral nerve block
  Interventions: Other: General anesthesia femoral continuous
- General anesthesia Femoral bolus (Active Comparator): General anesthesia plus single shot femoral nerve block
  Interventions: Other: General Anesthesia femoral bolus
- Femoral Sciatic Obturator Nerve block (Active Comparator): Ultrasound guided femoral plus sciatic plus obturator nerve block
  Interventions: Other: Ultrasound Guided Femoral Sciatic Obturator nerve blocks

INTERVENTIONS:
Other: Ultrasound Guided Femoral Sciatic Obturator nerve blocks
  Arms: Femoral Sciatic Obturator Nerve block
Other: General Anesthesia femoral bolus
  Arms: General anesthesia Femoral bolus
Other: General anesthesia femoral continuous
  Arms: General Anesthesia Femoral continuous

SUMMARY:
Arthroscopic ACL repair can be performed under different types of anesthesia. In the last few years peripheral nerve blocks have increased their popularity for this kind of operation. The investigators want to see how the type of anesthesia and postoperative analgesia effects the time required for patient mobilisation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 yrs
* ASA I - III
* ACL surgery

Exclusion Criteria:

* Coagulopathy disorders
* Infection at the puncture site for the interscalene block
* Neurologic deficit in the arm that is going to be operated
* Allergy to local anesthetics
* BMI > 35
* Psychiatric disorders
* Patient's refusal
* Problems with patient communication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Surgery completed without pain for the patient | Completion of the surgery
  Use of VAS score
Postoperative pain | 1st postoperative day
  Use of VAS score

SECONDARY OUTCOMES:
Mobilization of the knee | 24 weeks postoperatively
  How many degrees can the patient bend the knee

OTHER OUTCOMES:
Chronic pain development | 24 weeks postoperatively
  Use of questionnaire for the functional state of the knee and VAS score for the pain

CONTACTS AND LOCATIONS:
Overall Officials: Marina Simaioforidou, Medicine, Study Director — Private Clinic of Larissa "Asklipeiio"; George Basdekis, Medicine, Study Chair — Private Clinic of Larissa "Asklipeiio"; Konstantinos Bargiotas, Medicine, Study Chair — Larissa University Hospital; Aristeidis Zibis, Medicine, Study Chair — Private Clinic of Larissa "Askipeiio"; Athanasios Drakos, Medicine, Study Chair — Larissa University Hospital; Metaxia Bareka, Medicine, Principal Investigator — Larissa University Hospital
Locations (1):
- Private Clinic of Larissa "Asklipeiio", Larissa, Larissa, Greece